CLINICAL TRIAL: NCT02231099
Title: A Prospective and Comparative Study of the (Cost)Effectiveness Preformance of Tension Free Vaginal Mesh Plus Monocryl (Prolift+M) Versus Conventional Vaginal Prolaps Surgery in Primary Pelvic Organ Prolapse
Brief Title: Effectiveness Prolift+M Versus Conventional Vaginal Prolapse Surgery
Acronym: VROUW2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Principal Investigator, Mariella Withagen, Dr. M.I.J. Withagen, Radboud University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VROUW2
Record Dates: First submitted 2012-01-27; First posted 2014-09-04 (Estimated); Last update posted 2015-02-06 (Estimated); Status verified 2015-02

CONDITIONS: Pelvic Organ Prolapse; Cystocele; Rectocele; Uterine Prolapse
Keywords: recurrent pelvic organ prolapse; mesh
MeSH Terms: conditions — Pelvic Organ Prolapse; Cystocele; Rectocele; Uterine Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- prolift + m (Experimental): surgery with mesh (prolift+M)
  Interventions: Procedure: Prolift + M
- conventional vaginal prolapse surgery (Active Comparator): conventional vaginal prolapse surgery; anterior colporrhaphy or posterior colporrhaphy or spinal ligament fixation
  Interventions: Procedure: conventional vaginal prolapse surgery

INTERVENTIONS:
Procedure: Prolift + M — prolapse surgery with mesh
  Arms: prolift + m
Procedure: conventional vaginal prolapse surgery — conventional vaginal prolapse surgery;anterior colporrhaphy, posterior colporrhaphy
  Other Names: anterior colporrhaphy, posterior colporrhaphy
  Arms: conventional vaginal prolapse surgery

SUMMARY:
Pelvic organ prolapse is highly prevalent in the female population. The recurrence rate of pelvic organ prolapse after surgical treatment is high. This emphasizes the clinical need for improvement of the surgical techniques currently used. Placement of a mesh aims at reducing the recurrence rate.

In this study the investigators compare the effectiveness of the Tension free Vaginal mesh + Monocryl with standard vaginal prolapse surgery without mesh.

DETAILED DESCRIPTION:
Rationale: Pelvic organ prolapse is highly prevalent in the female population. The incidence of pelvic organ prolapse increases with age, so the longer life expectancy of women may cause pelvic organ prolapse to become an even more major health issue. The recurrence rate of pelvic organ prolapse after surgical treatment is high. The recurrence rate of the anterior vaginal wall prolapse after an anterior colporrhaphy is 30%-45%. The posterior vaginal wall prolapse recurrence rate after a posterior colporrhaphy is 12-25%. This emphasizes the clinical need for improvement of the surgical techniques currently used. Placement of a mesh aims at reducing the recurrence rate (2-11%).

Objective: To compare the clinical and cost effectiveness of the Tension free Vaginal Mesh + Monocryl (Prolift+M) with the standard vaginal prolapse surgery (i.e. fascial placation). A secondary objective is to track the post-operative and long-term complications of both procedures. A third objective is to evaluate recovery after surgery.

Study design: a prospective, multicentre, randomized, non-blinded study between Tension free Vaginal Mesh + Monocryl (Prolift+MTM) and standard vaginal prolapse surgery (i.e. fascial placation).

Study population: women with a primary pelvic organ prolapse of the anterior and/or posterior compartment POP stage II or more, in the age of 45 years or older.

Intervention (if applicable): Prolapse surgery with tension free vaginal mesh + Monocryl (Prolift + M) versus conventional vaginal prolapse surgery.

Main study parameters/endpoints: The main outcome is the percentage of patients with objective anatomical success (POP stage < 2) after 24 months. As secondary outcome the subjective improvement in quality of life will be measured by generic (EQ-5D,PGI-I) and disease-specific (UDI, DDI, IIQ and PFDI20) quality of life instrument. Sexual functioning will be measured by generic (FSFI) and disease specific (PISQ12) questionnaires. Complications will be monitored with special notice for pain (Mc Gill pain questionnaire) Recovery will be measured with the Recovery index 10. The economical endpoint is short term (2 year) incremental cost-effectiveness in terms of costs per additional year free of prolapse and costs per QALY gained.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Burden associated with participation: complete a disease specific Quality of life questionnaire 4 times, complete a recovery index questionnaire 3 times. Visit the hospital 4 times after the surgery (this is 2 times more often than patients not participating in the study). Since subjects are selected from subjects already agreeing to complete a surgical procedure, the additional risks of participation in this study are low. These risks include tissue erosion (vaginal, rectal or bladder), vaginal pain/dyspareunia.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a anterior and/or posterior prolapse POP-Q stage II or more. Subjects with a middle compartment prolapse may only be included if there is a co-existing anterior or posterior defect which needs surgical correction.
* Subject has agreed to undergo implantation of Prolift+MTM or fascial plication
* Subject is willing to return for follow-up evaluation and QoL questionnaires completion at 6weeks, 6 months, 12 months and 24 months follow-ups.

Exclusion Criteria:

* Pregnancy
* Age < 45 years
* Subject has had a previous surgery for pelvic organ prolapse. A previous mid-urethral sling procedure is not an exclusion criterion.
* Have current urinary tract or vaginal infections
* Have blood coagulation disorders
* Have a compromised immune system or any other conditions that would compromise healing
* Are unwilling or unable to return for evaluation
* Previous irradiation
* Presence of any malignancy

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2011-01; Primary Completion 2015-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
objective anatomic success (POPQ stage <2) | 24 months
  clinical investigation including POPQ

SECONDARY OUTCOMES:
subjective improvement in quality of life | 24 months
  Questionnaires; Euroqol5D, PGI-I, UDI, DDI and PFDI20
sexual function/dysfunction | 24 months
  PISQ-12, BESAQ
complications | 24 months
  clinical investigation
recovery | 6 weeks
  Recovery Index 10
cost-effectiveness | 24 months
  Costs of the strategies Tension free Vaginal mesh+Monocryl as well as standard vaginal prolapse surgery will be estimated using direct medical costs based on the actual costs of the surgery, personnel, material costs and costs for surgery due to recurrence or complications.

CONTACTS AND LOCATIONS:
Overall Officials: Mariella IJ Withagen, MD, PhD, Principal Investigator — Radboud Medical Center
Locations (5):
- Netherlands (5):
  - Gelre ziekenhuizen Apeldoorn, Apeldoorn
  - Reinier de Graaf Group, Delft
  - UMC St Radboud, Nijmegen
  - Zaans Medisch Centre, Zaandam
  - Isala clinics, Zwolle